CLINICAL TRIAL: NCT00383097
Title: Administration of LMP1- and LMP2- Specific Cytotoxic T-Lymphocytes Following CD45 Antibody to Patients With Relapsed EBV-Positive Hodgkin's or Non-Hodgkin's Lymphoma or Chronic Active EBV Infection (ALDI)
Brief Title: Lmp1 and Lmp2 Specific CTLs Following Cd45 Antibody for Relapsed Ebv-Positive Hodgkin's Or Non-Hodgkin's Lymphoma
Acronym: ALDI
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was terminated in 2010 due to lack of enrollment.
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Stephen Gottschalk, Principal Investigator, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19275; ALDI; NCT00608478 (obsolete NCT alias)
Record Dates: First submitted 2006-09-28; First posted 2006-10-02 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Hodgkins Lymphoma; Non-Hodgkin Lymphoma
Keywords: CTLs; LMP1; LMP2; CYTOTOXIC T-LYMPHOCYTES; CD45; ANTIBODY; EBV-POSITIVE HODGKIN'S; NON-HODGKIN'S LYMPHOMA
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: LMP1 SPECIFIC CYTOTOXIC T-LYMPHOCYTES — 1 injection One of the following 4 dose levels: 2x 10^7 cells/m2, 1x 10^8 cells/m2, 3 x 10^8 cells/m2, 1 x 10^9 cells/m2
Genetic: LMP2-SPECIFIC CYTOTOXIC T-LYMPHOCYTES — 1 injection One of the following 4 dose levels: 2x 10^7 cells/m2, 1x 10^8 cells/m2, 3 x 10^8 cells/m2, 1 x 10^9 cells/m2

SUMMARY:
The purpose of this study is to obtain blood (up to 90 ml or 18-teaspoonfuls on one or two occasions) to make LMP1- and LMP2-cytotoxic T-lymphocytes and grow them in the laboratory in such a way that they are able to attack LMP1- and LMP2-positive cells in the laboratory.

If we are successful in growing these cells and if we feel they would be helpful to the donor, we would then give the cells back to the donor.

This trial is for patients that have a type of lymph gland cancer called Hodgkin or non-Hodgkin lymphoma, or chronic active Epstein Barr virus (EBV) infection, which has come back or not gone away after treatment, including the best treatment we know.

This is a research study using special immune system cells called LMP1- and LMP2-specific cytotoxic T lymphocytes (LMP1- and LMP2-CTLs), a new experimental therapy. As in chronic active EBV infection, some patients with Hodgkin or non-Hodgkin lymphoma show evidence of infection with the virus that causes infectious mononucleosis (EBV) before or at the time of their diagnosis of the Lymphoma. EBV is found in the cancer cells of up to half the patients with lymphoma, suggesting that it may play a role in causing lymphoma. The cancer cells infected by EBV are able to hide from the body's immune system and escape destruction. We want to see if special white blood cells, called T cells, that have been trained to kill EBV infected cells can survive in the patient's blood and affect EBV-positive cells. In this present study we are trying to find out if we can improve this treatment by growing T cells that only recognize two of the proteins expressed on lymphoma cells called LMP1 and LMP2. These special T cells are called LMP1- and LMP2-specific cytotoxic CTLs.

DETAILED DESCRIPTION:
Infusions of CD45 MAbs A fixed dose of CD45 MAbs will be used determined from our previous and ongoing studies in stem cell transplant recipients will be used 40, 400ug/kg over 6 to 8 hrs daily x 4 given as daily intravenous infusions that will be completed 48-72 hours prior to CTL infusion. Patients will be premedicated prior to CD45 infusions and monitored as per the SOP for CD45 MAbs infusion.

Day 1 through Day 4: YTH 24/54 400ug/kg over 6 to 8 hr; Day 5: Rest; Day 6, 7 or 8: CTL Infusion (provided CD45 Mab level <100 ng/ml)

Preparation of the Patient:

Oxygen and suction equipment must be available in the room. Emergency drugs (Benadryl, Epinephrine, solucortef to solumedrol) in appropriate doses must be preordered by the physician prior to initiation of each infusion with doses available. A code card containing the appropriate doses of each medicine according to the patient's weight will also be available. Continuous telemetric monitoring by pulse oximeter and EKG will begin prior to and for 6 hours after each antibody infusion has taken place. Baseline vital signs are taken and recorded and monitored as per the SOP for antibody infusions.

MAbs Infusion:

The antibody aliquot to be infused will arrive in the treatment area hand-carried by the attending physician or appointed designate.

The antibody aliquot will be diluted in minimal amounts of normal saline. The resulting solution is stable for 24 hours.

The antibody solution is administered by a syringe pump in incremental doses, 0.2-0.8 mg in the first hour and up to 10 mg/hr thereafter, for a maximum infusion time of 8 hrs. A registered nurse and a physician must be readily available

Antibody toxicity:

Volume Overload: This is of particular importance in small recipients and will be monitored carefully.

Inflammatory mediator release from damaged circulating white cells and allergic reactions: Fever, chills, rigors, pruritis, urticaria, nausea, vomiting, throat tightness and dyspnea may occur. These reactions usually respond to slowing or stopping the infusion and/or the parenteral administration of diphenhydramine, hydrocortisone, meperidine or anti-emetics. Administration of O2, epinephrine, bronchodilators or IPPB may be necessary.

Adverse effects of CD45 MAbs on CTL Our experience to date has shown rapid clearance of CD45 MAbs from the plasma, such that levels are undetectable by 24-48hrs after infusion. However, the MAb levels will be measured before CTL infusion and if free plasma CD45 MAbs are present CTL infusion will be deferred for 24 hours

CTL Infusion:

Dose Levels of CTLs: The following dose levels will be evaluated: Each patient will receive 1 injection, according to the following dosing schedules:

Dose level I: 2 x 10e7 cells/m2; Dose level II: 1 x 10e8 cells/m2; Dose level III: 3 x 10e8 cells/m2; Dose level IV: 1 x 10e9 cells/m2. Patients will be pre-medicated with Benadryl 1mg/kg IV (max 50mg) and Tylenol 10mg/kg po (max 650mg).

Cell Administration: LMP1- and LMP2-specific T cells will be given by intravenous injection over 1-10 minutes through either a peripheral or a central line.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of EBV-positive Hodgkin's disease (HD), non-Hodgkin's lymphoma (NHL; all histological subtypes except Burkitt's lymphoma), or EBV (associated)-T/NK-LPD, or chronic active EBV infection (CAEBV) after second or subsequent relapse including after autologous or syngeneic stem cell transplant (or first relapse or with active disease if immunosuppressive chemotherapy contraindicated). CAEBV is defined as i) illness for greater than 3 months duration (EBV-related illness or symptoms including fever, persistent hepatitis, extensive lymphadenopathy, or hepatosplenomegaly); ii) increased amounts of EBV-DNA in peripheral blood (equal or greater than 400 genome copies per ug of DNA) or abnormal high levels of EBV antibodies (VCA IgG equal or greater than 1:5120 or EA IgG equal or greater than 1:640; and iii) no evidence of previous immunological abnormalities or other recent infection that might explain the observed condition.

Patients with life expectancy greater than 6 weeks.

Patients with a Karnofsky score (age ≥16) of greater than 50 or Lansky score (age<16) of greater than 50

No severe intercurrent infection.

HIV negative donor (if autologous donor, patient must be HIV negative)

Patient, parent/guardian able to give informed consent.

Patients with bilirubin less than3 x normal, AST less than 5 x normal, and Hgb greater than 8.0

Patients with a creatinine less than 2 x normal for age

Patients should have been off other investigational therapy including T cell therapies for one month prior to entry in this study.

Female patients with reproductive capacity must have a negative pregnancy test. Women of childbearing potential must not be pregnant and must be on effective birth control. The male partner should use a condom.

Note: Patients who would be excluded from the protocol strictly for laboratory abnormalities can be included at the investigator¡¦s discretion after approval by the CAGT Protocol Review Committee and the FDA reviewer.

Exclusion Criteria:

* Patient, parent/guardian unable or unwilling to give informed consent
* Pregnant women
* Patients with a Karnofsky score of < 50
* Patients with a severe intercurrent infection
* Patients with a life expectancy of <6 weeks
* Patients with a bilirubin greater than 3x normal. AST greater than 5x normal and Hgb less than 8.0 g/dl
* Patients with a creatinine greater than 2x normal for age
* Due to unknown effects of this therapy on a fetus, pregnant women are excluded from this research. The male partner should use a condom.

Note: Patients who would be excluded from the protocol strictly for laboratory abnormalities can be included at the investigator's discretion after approval by the CCGT Protocol Review Committee and the FDA reviewer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Dose limiting Toxicity: Two patients in each cohort are followed | 6 weeks post CTL infusion
Safety: All patients who received CD45 MAbs and LMP1- and LMP2-CTL infusions will be included in the safety analysis of this combination regimen | 1 year

SECONDARY OUTCOMES:
Laboratory data which includes CBC, BUN, creatinine, etc. will be examined at pre-infusion, and at 1, 2, 4, 6, 8 weeks post- CTL infusion, 3-month intervals for the first year | 1 year
Frequency of T cells specific for LMP1-, LMP2-, and other EBV-antigens as well as T cell specific for CMVpp65 will be measured and summarized at pre and post-infusion time points | 1 year
Changes of T cells specific for LMP1-, LMP2-, and other EBV-antigens as well as for CMVpp65 from pre-infusion to each time point of post-infusion in the overall patient group. | 1 year
Analysis of immunologic function of tetramer-positive cells in peripheral blood, and EBV-DNA in plasma will be performed at each time point of follow-up and paired comparisons of changes from baseline will be performed. | 1 year
Frequency of T cells specific for adenovirus and EBV. | 1 year
Analysis of anti-tumor activity; Overall response rates as well as by dose groups will be presented after the end of CTL infusion. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MALCOLM K BRENNER, MD, Study Director — Center for Cell and Gene Therapy, Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas